CLINICAL TRIAL: NCT04887532
Title: Safety and Pharmacokinetics of HR19042 Capsule After Single Administration in Healthy Chinese Subjects
Brief Title: A Trial of HR19042 Capsule in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HR19042-101
Record Dates: First submitted 2021-05-13; First posted 2021-05-14 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-05

CONDITIONS: Primary IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Intervention Model Description: Single center, open, three-period, sequential design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HR19042 capsule (Experimental)
  Interventions: Drug: HR19042 capsule

INTERVENTIONS:
Drug: HR19042 capsule — phase 1 :8mg; phase 2:12mg; phase 3:16mg

SUMMARY:
The study is being conducted to evaluate the safety and pharmacokinetics of HR19042 capsule after single administration in healthy Chinese subjects. To explore the pharmacokinetic characteristics and safety of HR19042 capsule in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 ~ 45 years old, including boundary value;
2. Female subjects weigh ≥45kg, male subjects weigh ≥50kg, and body mass index (BMI) is within the range of 19.0~26.0kg/m2 (body mass index = weight (kg)/height 2 (m2)), including boundary values;
3. The subject has no plans to give birth or donate sperm/eggs for at least 3 months from the signing of the informed consent form to the end of the study, and voluntarily take effective non-drug contraceptive measures (including partners) during the trial period;
4. Before the test, learn more about the nature, significance, possible benefits, possible inconvenience and potential risks of the test. Able to understand the procedures and methods of this research, willing to strictly abide by the clinical trial protocol to complete the trial, and voluntarily sign an informed consent form.

Exclusion Criteria:

1. People with a known history of drug or food allergies;
2. Past or current history of any disease that may affect the safety of subjects participating in the trial or the internal process of the research drug, including: digestive system, blood system, circulatory system, urinary system, respiratory system, nervous system, immune system, endocrine system, Those with a clear history of mental disorders and metabolic disorders, or other diseases that are not suitable for participating in clinical trials;
3. Those who have used drugs that affect the function of liver metabolic enzyme CYP3A4 within 30 days before the first administration (such as inducers-enzalutamide, mitotane, carbamazepine, phenytoin, rifampin; inhibitors-clarithromycin, irradian) Traconazole, ketoconazole, ritonavir, telithromycin, etc.), or those who have used contraceptives within 30 days before administration;
4. Those who have used any drug within 14 days before the first dose;
5. Those who have taken a special diet (including grapefruit/grapefruit juice, chocolate, food or beverages containing caffeine) within 48 hours before the first administration, or have consumed excessive amounts of tea, coffee or beverages containing caffeine every day for the past 1 month (Average more than 8 cups per day, 200 mL per cup);
6. Participate in drug clinical trials and take trial drugs as subjects within 3 months before screening, or plan to participate in other clinical trials during the study period;
7. Those who donated blood or lost more than 400 mL (excluding menstrual blood loss in women) within 3 months before screening, received blood transfusion or used blood products, or planned to donate blood during the trial period or within 1 month after the end of the trial;
8. Those who have undergone major surgery within 3 months before screening, or plan to undergo surgery during the study period;
9. Those who smoked more than 5 cigarettes a day on average in the 3 months before screening, or who did not agree to ban smoking during the trial;
10. In the 6 months before screening, the average weekly alcohol consumption exceeded 14 units of alcohol (1 unit = 360 mL of beer with 5% alcohol content or 45 mL of spirits with 40% alcohol content or 150 mL of wine with 12% alcohol content), Or those who do not agree to abstain from alcohol during the trial;
11. The results of laboratory tests (blood routine, urine routine, blood biochemistry, blood coagulation function) are judged by clinicians as abnormal and clinically significant;
12. Those whose 12-lead ECG, physical examination or vital signs examination results are judged by clinicians as abnormal and clinically meaningful;
13. Immunological examinations (hepatitis B surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, Treponema pallidum antibody) are positive;
14. Those with abnormal chest radiograph (posterior anterior position) and clinical significance;
15. Women who are pregnant or breastfeeding;
16. Those who have a positive alcohol breath test;
17. Those who have a positive urine drug screening;
18. Those who have a history of drug abuse or drug abuse;
19. People with a history of difficulty in venous blood collection, intolerance to venipuncture, or a history of fainting needles
20. Those who have difficulty swallowing, or have special dietary requirements and cannot follow a uniform diet;
21. The investigator believes that the subject has any other factors that are not suitable for participating in this trial (such as inability to understand the research requirements, poor compliance, infirmity, etc.).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-24 hours
  Peak concentration of drug observed from 0 hour to 24 hours after administration
AUC0-t; | 0-24 hours
  The area under the drug concentration-time curve at the sample collection time t that can be accurately determined from 0 hour to 24 hours after administration
AUC0-∞ | 0 hour to 24 hours
  The area under the concentration-time curve of drug from 0 hour to infinity after administration

SECONDARY OUTCOMES:
AE | Screening period to end of follow-up period, approximately 1 month
  Adverse event
the change of blood cortisol AUC0-24h from baseline after each cycle of administration | 0-24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China